CLINICAL TRIAL: NCT06547320
Title: Sensor-based Just-in Time Adaptive Interventions (JITAIs) Targeting Eating Behavior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DK122473 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Just-in-time Adaptive Intervention (Experimental): A sensor device called an Automatic Ingestion Monitor (AIM) will be worn on eyeglasses to monitor eating. Information from the device will be used to send messages to a smartphone to change eating behavior.
  Interventions: Behavioral: Eat Less Intervention; Behavioral: Eat Slower Intervention

INTERVENTIONS:
Behavioral: Eat Less Intervention — A sensor worn on eyeglasses monitors eating and provides messages to a smartphone when eating occurs to prompt small reductions in the amount of food eaten.
Behavioral: Eat Slower Intervention — A sensor worn on eyeglasses monitors eating and provides messages to a smartphone when eating occurs to prompt small reductions in the rate of eating.

SUMMARY:
The purpose of this study is to determine whether a sensor device called an Automatic Ingestion Monitor (AIM) that is worn on eyeglasses can be used with a smartphone to change eating behavior. Participants will wear the device for one week of no-intervention observation. They will then test behavioral interventions focused on eating for two weeks. The researchers hypothesize that messages sent to a smartphone that are based on information from the AIM can reduce the amount of food that is eaten and slow eating.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 27 and 45 kg/m-squared
* Weight stable within 5% in the past 6 months
* Self-reports basic familiarity with use of a smartphone

Exclusion Criteria:

* Diagnosed diabetes (type 1 and 2)
* Any poorly controlled medical condition that could affect weight and/or eating behavior (e.g., hypothyroidism)
* Medical conditions or use of medications or diets/supplements known to affect energy regulation or appetite
* Difficulty chewing or swallowing
* Diagnosed eating disorder
* Night or shift work
* Current participation in a weight loss program
* History of bariatric surgery
* Current pregnancy or lactation within the past 1 year, or planning a pregnancy during the study participation period
* Consuming a medically-prescribed or unusual diet (e.g., macrobiotic)
* Food allergies or sensitivities, or other conditions which result in avoidance of a wide range of foods (e.g. celiac disease, tree nut allergy)
* Reported recreational drug use
* Report of conditions that would significantly interfere with an ability to follow the protocol including terminal illness, substance abuse, or other significant uncontrolled psychiatric problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Total energy intake | Daily average computed for the 7-day observation period and each 7-day intervention period
  Total amount of energy consumed from foods and beverages

SECONDARY OUTCOMES:
Energy intake per eating occasion | Average intake per eating occasion computed for the 7-day observation period and each 7-day intervention period
  Amount of energy consumed from foods and beverages during each eating occasion
Rate of eating per eating occasion | Average intake per eating occasion computed for the 7-day observation period and each 7-day intervention period
  Chews per minute during each eating occasion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Boston University, Boston, Massachusetts
  - The Miriam Hospital Weight Control and Diabetes Resarch Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
We will make data and documentation available under a data-sharing agreement that provides for (1) a commitment to use the data for research purposes only; (2) a commitment to securing the data using appropriate computer technology; (3) a commitment to destroying or returning the data after analyses are completed and (4) a commitment not to attempt to identify participants individually. Information shared with outside collaborators will link personal health information to a unique study ID in order to maintain participant anonymity.
Supporting Information: Study Protocol, ICF
Access Criteria: A data-sharing agreement that provides for (1) a commitment to use the data for research purposes only; (2) a commitment to securing the data using appropriate computer technology; (3) a commitment to destroying or returning the data after analyses are completed and (4) a commitment not to attempt to identify participants individually. Information shared with outside collaborators will link personal health information to a unique study ID in order to maintain participant anonymity.